CLINICAL TRIAL: NCT02002494
Title: Effect of Different Surgical Positions on the Cerebral Venous Drainage: an Ultrasound Study on Healthy Volunteers
Brief Title: Jugular Venous Flow Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Lashmi Venkatraghavan, Dr., University Health Network, Toronto
Other Study IDs: 13-6244-BE
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Jugular Venous Blood Flow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- volunteers in different positions: The following will be compared in the same volunteer:
  * Bilateral internal jugular venous flow in supine and prone position
  * Bilateral internal jugular venous flow in supine and park bench position
  * Bilateral internal jugular venous flow in prone and park bench
  Interventions: Other: Different positions

INTERVENTIONS:
Other: Different positions — Jugular venous blood flow in healthy volunteers in 3 different positions- supine, prone and park bench

SUMMARY:
Our hypothesis is that there will be a decrease in internal jugular venous flow in the park bench position when compared to the supine position. There will also be a change in blood flow in the between right and left internal jugular veins in park bench position, particularly there will be a greater reduction of flow on the dependent side. However, the internal jugular venous flow will be the same in both the prone and supine position.

DETAILED DESCRIPTION:
The different positions used in neurosurgery (park bench, prone) for better accessibility to the operating field can impact on the cerebral venous drainage due to the effects of internal jugular venous outflow of blood and may increase intracranial pressure. The kinking of the internal jugular vein due to excessive neck flexion and rotation in park bench or flexion in the prone position may lead to kinking or twisting of the vein. This has been hypothesized as the major cause of disturbed venous drainage during surgery and in postoperative patients may lead to neck swelling, brachial plexus injury, macroglossia (swollen tongue), delayed airway obstruction and increases in intracranial pressure.

Optimal brain perfusion is best in the neutral position of the head, but surgery cannot always be performed with this. Thus, we look to measure the internal jugular venous flow at different positions as there have been little studies looking at this important contributing factor.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers who are above the age of 18
* American Society of Anesthesiologists classification (ASA) 1
* Body mass index (BMI) less than and equal to 35

Exclusion Criteria:

* ASA 2 and above
* BMI above 35
* Lack of informed consent
* Language barrier
* Medical students and anaesthesia residents going through the department as part of their rotation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lashmi Venkatraghavan, Principal Investigator — University Health Network, Toronto Western Hospital; Vincent Chan, Principal Investigator — University Health Network, Toronto Western Hospital; Pirjo Manninen, Principal Investigator — University Health Network, Toronto Western Hospital; Audrey MY Tan, Principal Investigator — University Health Network, Toronto Western Hospital
Locations (1):
- University Health Network, Toronto Western Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-seven volunteers were included in this study.
Groups:
- Volunteers in Different Positions: The following will be compared in the same volunteer:
  * Bilateral internal jugular venous flow in supine and prone position
  * Bilateral internal jugular venous flow in supine and park bench position
  * Bilateral internal jugular venous flow in prone and park bench Different positions: Jugular venous blood flow in healthy volunteers in 3 different positions- supine, prone and park bench
Period: Overall Study
Arm/Group | Volunteers in Different Positions
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Twenty-seven volunteers were included in this study. The mean (SD) age, height and weight of these participants were analyzed.
Arm/Group | Volunteers in Different Positions
Number analyzed (Participants) | 27
Age, Customized [Mean (Standard Deviation); unit: years] | 38 (10)
Sex/Gender, Customized [Number; unit: participants] | 27
Height [Mean (Standard Deviation); unit: units on a scale] | 169.5 (12.5)
Weight [Mean (Standard Deviation); unit: units on a scale] | 71.8 (15.4)

OUTCOME MEASURES:

1. Primary Outcome: Internal Jugular Venous (IJV) Cross Sectional Area
Description: Comparisons of both jugular vein (IJV) of twenty-seven volunteers in supine and prone positions.
Time Frame: 1 day
Population: Twenty-seven volunteers were included in this study. Comparisons of right and left internal jugular vein (IJV) cross sectional area, Doppler velocity and flow between supine and prone position.
Measure: Mean (Standard Deviation); unit: cm2
Groups:
- R IJV: Comparisons of right internal jugular vein (IJV) cross sectional area, Doppler velocity and flow between supine and prone position.
- L IJV: Comparisons of left internal jugular vein (IJV) cross sectional area, Doppler velocity and flow between supine and prone position.
Arm/Group | R IJV | L IJV
Number analyzed (Participants) | 27 | 27
cm2
  Supine-Cross sectional area | 1.2 (0.6) | 1.0 (0.3)
  Prone-Cross sectional area | 1.8 (1) | 1.4 (0.4)

2. Primary Outcome: Right and Left IJV Cross Sectional Area
Description: Twenty-seven volunteers were included in this study. Comparisons of cross sectional area measurements in both IJVs between supine and right park bench
Time Frame: 1 day
Population: Comparisons of bilateral internal jugular vein (IJV) cross sectional area, Doppler velocity and flow between supine and right park bench position.
Measure: Mean (Standard Deviation); unit: cm2
Groups:
- R IJV: - We studied R IJV flow in the supine and right park bench positions respectively.
  all measurements were performed on the right eye in a neutral gaze.
  - We standardised the use of the right side because of ease of access to that side in the laboratory.
- L IJV: - We studied L IJV flow in the supine and right park bench positions respectively.
  all measurements were performed on the right eye in a neutral gaze.
  - We standardised the use of the right side because of ease of access to that side in the laboratory.
Arm/Group | R IJV | L IJV
Number analyzed (Participants) | 27 | 27
cm2
  Supine-Cross sectional area (cm2) | 1.2 (0.6) | 1.0 (0.3)
  Right park bench-Cross sectional area | 0.9 (0.5) | 1.1 (0.5)

3. Primary Outcome: Internal Jugular Venous (IJV) Doppler Velocity
Description: 27 volunteers enrolled to measure the Internal Jugular Venous (IJV) in supine and prone positions
Time Frame: 1 day
Population: Comparisons of bilateral internal jugular vein (IJV) Doppler velocity between supine and prone position. Data presented as mean (SD) .
Measure: Mean (Standard Deviation); unit: cm.sec-1
Groups:
- R IJV: Comparisons of right internal jugular vein (IJV) Doppler velocity between supine and prone position.
- L IJV: Comparisons of left internal jugular vein (IJV) Doppler velocity between supine and prone position.
Arm/Group | R IJV | L IJV
Number analyzed (Participants) | 27 | 27
cm.sec-1
  Supine Doppler velocity | 19.9 (7) | 18.1 (8.4)
  Prone Doppler velocity | 19.3 (7.9) | 13.6 (7.7)

4. Primary Outcome: Bilateral Internal Jugular Vein (IJV) Flow
Description: Comparisons of bilateral internal jugular vein (IJV) flow between supine and prone position. Data presented as mean (SD) .
Time Frame: 1 day
Population: Comparisons of bilateral internal jugular vein (IJV) flow between supine and prone position. Data presented as mean (SD) .
Measure: Mean (Standard Deviation); unit: ml.min-1
Groups:
- R IJV: Comparisons of right internal jugular vein (IJV) flow between supine and prone position.
- L IJV: Comparisons of left internal jugular vein (IJV) flow between supine and prone position.
Arm/Group | R IJV | L IJV
Number analyzed (Participants) | 27 | 27
ml.min-1
  Supine Flow | 1430.1 (803) | 1112.9 (578.1)
  Prone Flow | 1924.2 (1139.7) | 1178.4 (832.1)

5. Primary Outcome: Bilateral Internal Jugular Vein (IJV) Doppler Velocity
Description: Comparisons of bilateral internal jugular vein (IJV) Doppler velocity between supine and right park bench position.
Time Frame: 1 day
Population: Comparisons of bilateral internal jugular vein (IJV) cross sectional area, Doppler velocity and flow between supine and right park bench position. Data presented as mean (SD).
Measure: Mean (Standard Deviation); unit: cm.sec-1
Groups:
- R IJV: Comparisons of right internal jugular vein (IJV) Doppler velocity between supine and right park bench position
- L IJV: Comparisons of left internal jugular vein (IJV) Doppler velocity between supine and right park bench position
Arm/Group | R IJV | L IJV
Number analyzed (Participants) | 27 | 27
cm.sec-1
  supine Doppler velocity | 19.9 (7) | 18.1 (8.4)
  right park bench Doppler velocity | 28.1 (12) | 18.7 (11.6)

6. Primary Outcome: R IJV and L IJV Flow
Description: Bilateral internal jugular vein (IJV) flow between supine and right park bench position.
Time Frame: 1 day
Population: Comparisons of bilateral internal jugular vein (IJV) flow between supine and right park bench position. Data presented as mean (SD).
Measure: Mean (Standard Deviation); unit: ml.min-1
Groups:
- R IJV: Comparisons of right internal jugular vein (IJV) Flow between supine and right park bench position
- L IJV: Comparisons of left internal jugular vein (IJV) Flow between supine and right park bench position
Arm/Group | R IJV | L IJV
Number analyzed (Participants) | 27 | 27
ml.min-1
  supine Flow | 1430.1 (803) | 1112.9 (578.1)
  right park bench Flow | 1403.1 (1006.1) | 1266.9 (959.6)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Volunteers in Different Positions
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes